CLINICAL TRIAL: NCT07030608
Title: The Effect of Pelvic Floor Muscle Exercises on Sexual Life in Women With Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Nezihe KIZILKAYA BEJI, Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/60-11
Record Dates: First submitted 2025-05-30; First posted 2025-06-22 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-06

CONDITIONS: Sexual Function; Over Active Bladder
Keywords: over active bladder; Pelvic Floor Muscle; sexual function
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study included 64 women admitted to the Erzurum City Hospital, who consented to participate. They were divided into intervention and controls groups (n=32). PFME (Pelvic Floor Muscle Exercise) was applied to the intervention group for 6 weeks with the Simplex Device accompanied by biofeedback in accordance with the PFME application procedure. The control group received routine care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Women in the control group did not receive any intervention or pelvic floor muscle exercise training.
- Intervention (Experimental): The intervention group performed a pelvic floor muscle exercise program in addition to the pharmacological treatment routinely provided at the hospital. Pelvic Floor Muscle Exercise Program Week 1: Contract the pelvic floor muscles for 6 seconds, then relax for 6 seconds. Repeat 25 times. Perform 3 sessions per day (total of 75 contractions per day). Week 2: Contract for 6 seconds, relax for 6 seconds. Repeat 50 times. Perform 3 sessions per day (total of 150 contractions per day). Week 3: Contract for 6 seconds, relax for 6 seconds. Repeat 75 times. Perform 3 sessions per day (total of 225 contractions per day). Weeks 4-24: Contract for 6 seconds, relax for 6 seconds. Repeat 100 times. Perform 3 sessions per day (total of 300 contractions per day). After Week 24: Contract for 6 seconds, relax for 6 seconds. Repeat 50 times. Perform 3 sessions per day (total of 150 contractions per day).
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Pelvic Floor Muscle Exercise Program Week 1: Contract the pelvic floor muscles for 6 seconds, then relax for 6 seconds. Repeat 25 times. Perform 3 sessions per day (total of 75 contractions per day). Week 2: Contract for 6 seconds, relax for 6 seconds. Repeat 50 times. Perform 3 sessions per day (total of 150 contractions per day). Week 3: Contract for 6 seconds, relax for 6 seconds. Repeat 75 times. Perform 3 sessions per day (total of 225 contractions per day). Weeks 4-24: Contract for 6 seconds, relax for 6 seconds. Repeat 100 times. Perform 3 sessions per day (total of 300 contractions per day). After Week 24: Contract for 6 seconds, relax for 6 seconds. Repeat 50 times. Perform 3 sessions per day (total of 150 contractions per day).
  Arms: Intervention

SUMMARY:
This is a randomized controlled experimental study to determine the effect of pelvic floor muscle exercise on sexual life.

The study included 64 women admitted to the Erzurum City Hospital, who consented to participate. They were divided into intervention ond control groups (n=32). Pelvic Floor Muscle Exercise *PFME* was applied to the intervention group for 6 weeks with the Simplex Device accompanied by biofeedback in accordance with the PFME application procedure. The control group received routine care.

DETAILED DESCRIPTION:
This is a randomized controlled experimental study . The research was carried out in the Erzurum City Hospital. This study, which was conducted to examine the effect of pelvic floor muscle exercises *PFME* on sexual life in women with overactive bladder *OAB* , was conducted with 64 women (32 women: control group, 32 women: intervention group) who applied to the Erzurum City Hospital Urology Polyclinic between December 1, 2021 and December 1, 2024.

Research Hypotheses:

H1: Overactive bladder symptoms are positively affected in women with OAB who perform pelvic floor exercises.

H2: Sexual function is positively affected in women with OAB who perform pelvic floor exercises.

H3: Depression symptoms are positively affected in women with OAB who perform pelvic floor exercises.

H4: Sexual quality of life is positively affected in women with OAB who perform pelvic floor exercises.

H5: Pelvic muscle strength increases in women with OAB who undergo pelvic floor muscle training.

H6: The contraction, relaxation, and percentage of maximum voluntary contraction *MVC* % of pelvic floor muscles improve in women with OAB who undergo pelvic floor muscle training.

Implementation:

The intervention group performed a pelvic floor muscle exercise program in addition to the pharmacological treatment routinely provided at the hospital. Pelvic floor muscle exercises-including identifying the correct muscle, contraction, and relaxation-were taught by the researcher using biofeedback via the Simplex device. The training was reinforced through the use of biofeedback techniques, including a game integrated into the Simplex software, as well as verbal cues provided by the researcher .

To ensure proper continuation of the exercises and to help participants remember them, a handbook prepared by the researcher was provided (Pelvic Floor Muscle Exercise Training Handbook for Women with Overactive Bladder). Participants were asked to complete the Pelvic Floor Muscle Exercise Practice Tracking Form after each exercise session.

Additionally, the women were contacted weekly by the researcher via telephone. They were either invited to the hospital for follow-up or visited at home for evaluation and feedback.

Pelvic Floor Muscle Exercise Program

Week 1:

Contract the pelvic floor muscles for 6 seconds, then relax for 6 seconds. Repeat 25 times. Perform 3 sessions per day (total of 75 contractions per day).

Week 2:

Contract for 6 seconds, relax for 6 seconds. Repeat 50 times. Perform 3 sessions per day (total of 150 contractions per day).

Week 3:

Contract for 6 seconds, relax for 6 seconds. Repeat 75 times. Perform 3 sessions per day (total of 225 contractions per day).

Weeks 4-24:

Contract for 6 seconds, relax for 6 seconds. Repeat 100 times. Perform 3 sessions per day (total of 300 contractions per day).

After Week 24:

Contract for 6 seconds, relax for 6 seconds. Repeat 50 times. Perform 3 sessions per day (total of 150 contractions per day).

Alternatively (preferred option):

Contract for 6 seconds, relax for 6 seconds. Repeat 75 times. Perform 2 sessions per day (total of 150 contractions per day).

Women in the control group did not receive any intervention or pelvic floor muscle exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 70 years of age
* Speaking Turkish
* Being literate
* Having a diagnosis of Overactive Bladder (OAB)
* Currently receiving pharmacological treatment for OAB
* Being willing to participate in the study voluntarily

Exclusion Criteria:

* Presence of perceptual impairments or psychiatric disorders that interfere with communication
* Diagnosis of a neurological disease
* Presence of neuropathy due to Diabetes Mellitus
* Pelvic organ prolapse at Stage 2 or higher
* History of anti-incontinence surgery
* Being pregnant

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Over active bladder questionnaire | Change from beginning of the study and after 6th week of exercise program
  This questionnaires evaluates urination frequency, sudden feeling of urgency, nocturia, urge type incontinence symptoms. It consists of 8 questions that patients can rate the severity of their complaints as none (0); very little (1); a little (2); quite a bit (3); a lot (4); and very much (5).
pelvic floor muscle contraction strength | Change from beginning of the study and after 6th week of exercise program
  Pelvic floor muscle strength measurement by digital palpation
pelvic floor muscle contraction strength | Change from beginning of the study and after 6th week of exercise program
  Pelvic floor muscle strength measurement by Simplex device
pelvic floor muscle relaxation strength | Change from beginning of the study and after 6th week of exercise program
  Pelvic floor muscle strength measurement by Simplex device
Female Sexual Function Index Scores ≤ 26.55 | Change from beginning of the study and after 6th week of exercises program
  The Female Sexual Function Index consists of 19 items that measure six domains of female sexual function:
  Desire (2 items)
  Arousal (4 items)
  Lubrication (4 items)
  Orgasm (3 items)
  Satisfaction (3 items)
  Pain (3 items; includes discomfort during or after vaginal penetration) Each item is scored on a Likert-type scale, typically ranging from 0 or 1 to 5.Total score range: 2.0 to 36.0 Cut-off score: A total FSFI score of ≤26.55 is commonly used to indicate female sexual dysfunction (FSD).
Center of Epidemiologic Studies Depression Scale | Change from beginning of the study and after 6th week of exercise program.
  The Center of Epidemiologic Studies Depression Scale is designed to assess the frequency and severity of symptoms associated with depression. The original CES-D contains 20 items.Each item is scored on a 4-point Likert scale:
  0 = Rarely or none of the time (<1 day)
  1. = Some or a little of the time (1-2 days)
  2. = Occasionally or a moderate amount of time (3-4 days)
  3. = Most or all of the time (5-7 days)
  Total scores range from 0 to 60.
  A score of 16 or higher is generally used as a cut-off to indicate significant levels of depressive symptoms, though this is not a diagnostic tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni Üniversitesi, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators did not obtain permission from the participants to share their data with other researchers.